CLINICAL TRIAL: NCT03445390
Title: The Effect of Intravenous Acetaminophen on Post-Operative Pain After Craniotomy: A Randomized Control Trial
Brief Title: The Effect of Intravenous Acetaminophen on Post-Operative Pain After Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Mark Burbridge, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 27467
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Patients selected for this study were being treated for Moyamoya disease and required two operations, scheduled 1-2 weeks apart. With random assignment, patients were administered 1 gram of intravenous acetaminophen at the beginning and end of surgery, and placebo during the other operation.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen First (Experimental): Patients in this group are presenting for 2 surgeries and will be administered intravenous acetaminophen in one surgery and placebo in the other. Patients in this group will be randomized to receive acetaminophen first.
  Interventions: Drug: Acetaminophen; Drug: Placebo
- Placebo First (Experimental): Patients in this group are presenting for 2 surgeries and will be administered intravenous acetaminophen in one surgery and placebo in the other. Patients in this group will be randomized to receive placebo first.
  Interventions: Drug: Acetaminophen; Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 1 g intravenous given at the beginning and end of surgery.
  Other Names: Tylenol
Drug: Placebo — Placebo to match acetaminophen given at the beginning and end of surgery.

SUMMARY:
The purpose of the study is to determine the efficacy of IV acetaminophen when administered to neurosurgical patients at the beginning and end of their surgery. If the result is improved pain control with less opioid consumption postoperatively, then those patients may also experience less opioid related side effects such as nausea/vomiting, pruritus, and sedation. While numerous other studies have failed to show a benefit of IV acetaminophen after neurosurgical procedures, we are studying the administration of 1 g in two doses over the course of the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of bilateral moyamoya disease scheduled for bilateral external-carotid to internal-carotid bypass surgery to be done in two stages.

Exclusion Criteria:

* Allergy or history of reaction to acetaminophen. Patients with liver disease. Anyone not able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen First, Then Placebo; Placebo First, Then Acetaminophen: Patients were administered intravenous acetaminophen (1 g IV) twice in one surgery and placebo to match in the other. Patients were randomly assigned to acetaminophen first or placebo first.
Period: First Intervention
Arm/Group | Acetaminophen First, Then Placebo | Placebo First, Then Acetaminophen
Started | 14 | 13
Completed | 12 | 11
Not Completed | 2 | 2
Period: Second Intervention
Arm/Group | Acetaminophen First, Then Placebo | Placebo First, Then Acetaminophen
Started | 12 | 11
Completed | 10 | 10
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed both interventions were included in the analysis.
Groups:
- All Study Participants: Patients were administered intravenous acetaminophen (1 g IV) twice in one surgery and placebo to match in the other. Patients were randomly assigned to acetaminophen first or placebo first.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Opioid Consumption
Description: From nursing records how much opioid was administered to each patient post-operatively. Opioid use was measured in micrograms (ug) of fentanyl.
Time Frame: Up to 24 hours post-operative
Population: Participants who completed both interventions were included in the analysis.
Measure: Mean (Standard Deviation); unit: ug
Groups:
- Acetaminophen: Patients were administered intravenous acetaminophen (1 g IV) twice.
- Placebo: Patients were administered placebo to match acetaminophen.
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 20 | 20
ug | 228 (125) | 312 (165)

2. Primary Outcome: Post-operative Pain
Description: Patients were asked to rate their pain on a scale of 1 to 10, with 1 being least pain, and 10 being most pain. Pain was assessed continually once per hour during the post-operative period and the average pain score calculated per participant. The average of the participants' average scores is presented for each group.
Time Frame: Up to 24 hours post-operative
Population: Participants who completed both interventions were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Post-operative hour 0 to 12 | 3.4 (2.6) | 3.8 (1.8)
  Post-operative hour 13 to 24 | 2.7 (2.5) | 2.6 (1.8)
  Post-operative hour 0 to 24 | 3.1 (2.4) | 3.2 (1.7)

3. Secondary Outcome: Count of Participants Requiring Anti-emetic Administration
Time Frame: Up to 24 hours post-operative
Population: Participants who completed both interventions were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

ADVERSE EVENTS:
Time Frame: Up to 2 weeks
Arm/Group | Acetaminophen | Placebo
All-Cause Mortality (participants affected / at risk) | 2/25 | 2/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2013-05-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT03445390/Prot_000.pdf